CLINICAL TRIAL: NCT07202013
Title: Clinical Evaluation of Kinesio Taping Outcomes in Stage II Cellulite: a Pilot Randomised Controlled Trial
Brief Title: Pilot Trial of Kinesio Taping in Stage II Cellulite
Acronym: CELLTAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klaipedos valstybine kolegija (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CELLULITE-KT-RCT-01; 2024-12-27, Nr. SSV6-114 (Other: Klaipedos valstybine kolegija/Higher Education Institution)
Record Dates: First submitted 2025-09-16; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cellulite of Thighs
Keywords: cellulite; Kinesio Taping; Skin Structure; Dermis Density; Low Echogenic Band; Body composition
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping (Experimental): Participants received kinesio taping once weekly for four weeks. Fan-shaped elastic therapeutic tape was applied with 0-15% tension to the thighs and buttocks, including the gluteus maximus, posterior thigh, and anterior thigh, to promote lymphatic drainage, improve microcirculation, and support skin structure.
  Interventions: Other: Kinesio taping
- No intervention (No Intervention): Participants in this arm did not receive any intervention during the study period. They completed the same baseline, post-intervention (4 weeks) assessments as the experimental group to allow comparison of outcomes without kinesio taping.

INTERVENTIONS:
Other: Kinesio taping — Kinesio taping was applied in a fan-shaped pattern once weekly for four consecutive weeks. Elastic therapeutic tape was applied with 0-15% tension to the buttocks and thighs at standardized anatomical points, including the gluteus maximus (above the sacroiliac joint), posterior thigh (gluteal fold), and anterior thigh (above the anterior inferior iliac crest). This protocol was designed to promote lymphatic drainage, improve microcirculation, and enhance dermal density and structure in women with stage II cellulite.
  Arms: Kinesio taping

SUMMARY:
The goal of this clinical trial is to evaluate whether kinesio taping can improve skin structure and reduce stage II cellulite in women. The study focuses on adult female participants aged 18-45 with stage II cellulite and normal BMI.

The main questions it aims to answer are:

Does kinesio taping increase dermis density? Does kinesio taping improve low echogenic band (LEB) thickness, an ultrasound marker of skin structure? Researchers will compare an experimental group receiving weekly fan-shaped kinesio tape applications on thighs and buttocks for four weeks to a control group that receives no intervention, to see if kinesio taping improves clinical and instrumental measures of cellulite.

Participants will:

Undergo baseline and follow-up assessments, including body composition, thigh circumference, cellulite stage scoring, and ultrasound of dermis density and LEB.

In the experimental group, receive kinesio taping applied once weekly for four weeks on the buttocks and thighs.

Return for re-evaluation immediately after the intervention and four weeks later.

DETAILED DESCRIPTION:
Cellulite is a common skin condition characterized by dimpling and irregular surface texture, primarily affecting women. It is associated with changes in the dermis and subcutaneous connective tissue, impaired microcirculation, and lymphatic congestion. Although not a disease, cellulite negatively impacts quality of life and has psychosocial consequences. Stage II cellulite, as defined by the Nürnberger-Müller Scale, presents with visible dimpling when standing, structural changes on palpation, and alterations detectable through imaging.

Kinesio taping (KT) is a non-invasive physiotherapy method widely used for musculoskeletal and circulatory conditions. Elastic tape is applied to the skin in specific patterns with the aim of lifting the epidermis, reducing local pressure, improving interstitial fluid flow, and enhancing lymphatic drainage. Based on these mechanisms, KT may be beneficial in the treatment of cellulite, particularly by improving dermal structure and promoting metabolic activity in subcutaneous fat. However, scientific evidence for KT in cellulite management remains scarce and inconsistent.

This pilot randomised controlled trial is designed to evaluate the short-term effects of kinesio taping on structural skin parameters in women with stage II cellulite. Thirty-four participants aged 18-45 years with normal body mass index and clinically confirmed stage II cellulite are randomly assigned to an experimental group or a control group. The experimental group receives fan-shaped kinesio tape applied once weekly for four weeks on the buttocks and thighs. The control group receives no intervention during the study period.

Primary outcomes include dermis density and low echogenic band (LEB) thickness measured using high-frequency ultrasound (DermaLab Combo 4). Secondary outcomes include cellulite stage scoring (Nürnberger-Müller Scale and Callegari Soft Plus), thigh circumference, body composition (fat percentage, fat mass, fat-free mass, basal metabolic rate, and total body water), and skin moisture. Measurements are taken at baseline, after four weeks of intervention, and four weeks post-intervention to assess residual effects.

The primary hypothesis is that kinesio taping will increase dermis density and LEB thickness compared with no intervention, indicating improved skin structure. Secondary hypotheses include potential reductions in thigh circumference and fat percentage and stabilization of skin hydration compared to the control group.

This study is exploratory and intended to provide pilot data on feasibility, effect sizes, and outcome variability. Findings may inform the design of larger trials and contribute to the evidence base for kinesio taping as a possible adjunctive therapy in cellulite management.

ELIGIBILITY:
Inclusion Criteria:

* women,
* aged 18-45,
* with Stage II cellulite,
* normal BMI

Exclusion Criteria:

* pregnancy,
* edema,
* obesity,
* thrombosis,
* skin infections

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Low Echogenic Band (LEB) Thickness | Baseline to 4 weeks (end of intervention).
  LEB thickness, a subepidermal ultrasound marker of skin integrity and cellulite severity, will be measured using high-frequency ultrasound (DermaLab Combo 4).
Change in Dermis Density | Baseline to 4 weeks (end of intervention).
  Dermis density will be assessed using high-frequency ultrasound (DermaLab Combo 4) to evaluate changes in skin structure associated with cellulite.

SECONDARY OUTCOMES:
Change in Thigh Circumference | Baseline to 4 weeks (end of intervention)
  Thigh circumference measured 20 cm below the greater trochanter with participants standing relaxed, to assess reduction in girth associated with cellulite.
Change in Body Fat Percentage | Baseline to 4 weeks (end of intervention)
  Body fat percentage will be measured by bioelectrical impedance analysis (Tanita BC-418MA).
Change in Cellulite Stage (Nürnberger-Müller Scale) | Baseline to 4 weeks (end of intervention)
  Cellulite severity will be assessed using the Nürnberger-Müller Scale. Minimum = 0 (no cellulite) Maximum = 3 (severe cellulite) Higher scores indicate worse cellulite severity. Higher scores indicate worse cellulite severity.
Change in Cellulite Severity (Callegari Soft Plus System) | Baseline to 4 weeks (end of intervention)
  Cellulite severity will be measured using the Callegari Soft Plus system, which provides a continuous numerical score based on skin tissue analysis.
  Minimum = 0 (no detectable cellulite) Maximum = 100 (severe cellulite).Higher scores indicate worse cellulite severity.
Change in Fat Mass (kg) | Baseline to 4 weeks (end of intervention)
  Fat mass will be measured by bioelectrical impedance analysis (Tanita BC-418MA).
Change in Fat-Free Mass (Kg) | Baseline to 4 weeks (end of intervention)
  Fat-free mass will be measured by bioelectrical impedance analysis (Tanita BC-418MA).
Change in Basal Metabolic Rate (kcal/day) | Baseline to 4 weeks (end of intervention)
  Basal metabolic rate will be measured by bioelectrical impedance analysis (Tanita BC-418MA).
Change in Total Body Water (%) | Baseline to 4 weeks (end of intervention)
  Total body water will be measured by bioelectrical impedance analysis (Tanita BC-418MA).

CONTACTS AND LOCATIONS:
Overall Officials: Laura Zaliene, PhD, Principal Investigator — Klaipedos valstybine kolegija
Locations (1):
- Klaipedos valstybine kolegija, Klaipėda, Lithuania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT07202013/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT07202013/SAP_001.pdf
  • Informed Consent Form (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT07202013/ICF_002.pdf